CLINICAL TRIAL: NCT02413242
Title: Advanced Understanding of Staphylococcus Aureus and Pseudomonas Aeruginosa Infections in EuRopE - ICU
Acronym: ASPIRE-ICU
Status: Completed | Type: Observational
Sponsor: Jan Kluytmans (Other)
Collaborators: MedImmune LLC (Industry); Universiteit Antwerpen (Other)
Responsible Party: Sponsor-Investigator, Jan Kluytmans, Professor, UMC Utrecht
Organization: UMC Utrecht (Other)
Other Study IDs: NL51762.041.14
Record Dates: First submitted 2015-04-01; First posted 2015-04-09 (Estimated); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Pneumonia; Pneumonia, Ventilator-Associated; Nosocomial Pneumonia
Keywords: S. aureus; P. aeruginosa; Colonization; Pneumonia; ICU
MeSH Terms: conditions — Pneumonia; Pneumonia, Ventilator-Associated; Healthcare-Associated Pneumonia; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Microbiological samples:
    * Nose swabs - at day of informed consent form (ICF), day 4, day 7.
    * Peri-anal swabs - at day of ICF, day 4, day 7, then twice weekly until day 30.
    * Lower respiratory tract (LRT) sample - at day of ICF, day 4, day 7, then twice weekly until day 30, day of ICU pneumonia, day 7 after ICU pneumonia. The LRT sample can be defined as the collection of an endotracheal aspirate (ETA). If an ETA cannot be collected, a sputum sample may be taken.
    * Broncho alveolar lavage - If available through clinical procedures, BAL specimens will be collected for study purposes.
  * Blood samples * Blood samples will be taken at day of ICF, day 7 and day 30 or day of ICU discharge (whichever occurs first), day of ICU pneumonia, day 7 after ICU pneumonia and day 30 after ICU pneumonia.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ICU subjects, S. aureus+ at ICU admission: Adult ICU patients, with a positive colonization status for S. aureus at ICU admission, who are mechanically ventilated within 24 hours of ICU admission and have an expected length of stay of 48h or more.
  Colonization status will be measured at ICU admission using a nose swab and an ETA (or sputum/throat if unavailable). Positivity of either of the two qualifies the patient to be enrolled as a subject in this group.
  Interventions: Other: Various observed exposure(s) of interest
- ICU subjects, S. aureus- at ICU admission: Adult ICU patients, with a negative colonization status for S. aureus at ICU admission, who are mechanically ventilated within 24 hours of ICU admission and have an expected length of stay of 48h or more.
  Colonization status will be measured at ICU admission using a nose swab and an ETA (or sputum/throat if unavailable). Negativity of both qualifies the patient to be enrolled as a subject in this group.
  Interventions: Other: Various observed exposure(s) of interest

INTERVENTIONS:
Other: Various observed exposure(s) of interest — A risk prediction model will be developed to assess which risk factors are associated with the development of ICU pneumonia during ICU stay

SUMMARY:
Intensive Care Unit (ICU) acquired pneumonia, including ventilator-associated pneumonia, is a frequently occurring health-care associated infection, which causes considerable morbidity, mortality and health care costs. Important pathogens causing ICU pneumonia are Staphylococcus aureus and Pseudomonas aeruginosa. The epidemiology of ICU pneumonia and patient-related and contextual factors is not fully described, but is urgently needed to support the development of effective interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is 18 years or older at the time of enrollment.
2. Participant is on mechanical ventilation at ICU admission, or is (expected to be) within 24 hours thereafter, based on investigator's judgment.
3. Expected stay in ICU is 48 hours or longer based on investigator's judgment.
4. SA colonization status is known within 72 hours after start of first episode of mechanical ventilation and according to the result, the patient qualifies for enrollment.
5. Written informed consent from subject / legally accepted representative within 72 hours after start of first episode of mechanical ventilation.

Exclusion Criteria:

1. Previous participation as a subject in the study cohort of this study.
2. Simultaneous participation of the subject in any preventive experimental study into anti-staphylococcus or anti-pseudomonas aeruginosa interventions.
3. Expected death (moribund status) within 48h, or ICU discharge of the participant within 24h, at the moment of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients in approximately 30 sites in 6-12 European countries will be selected based on eligibility criteria that are described below.
  Inclusion will be based on S. aureus (SA) colonization status at ICU admission (ratio 1:1). These subjects will be followed through their ICU stay for assessment of the primary outcomes.
Sampling Method: Probability Sample
Enrollment: 2031 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of S. aureus ICU pneumonia | date of ICF until ICU discharge (on average 7 days after ICF)
Incidence of P. aeruginosa ICU pneumonia | date of ICF until ICU discharge (on average 7 days after ICF)

SECONDARY OUTCOMES:
Prevalence of S. aureus / P. aeruginosa colonization | at ICU admission
Incidence of all cause ICU pneumonia | date of ICF until ICU discharge (on average 7 days after ICF)
Incidence of S. aureus ICU pneumonia stratified by MRSA vs. MSSA | date of ICF until ICU discharge (on average 7 days after ICF)
Incidence of P. aeruginosa ICU pneumonia stratified by MDR-PA vs. S-PA | date of ICF until ICU discharge (on average 7 days after ICF)
Incidence of ICU bacteremia per etiologic agent (in case of S. aureus and/or P. aeruginosa and for all clinically relevant other pathogens) | date of ICF until ICU discharge (on average 7 days after ICF)
All-cause mortality | date of ICF until ICU discharge (on average 7 days after ICF)
All-cause mortality | At day 30 after ICU admission
All-cause mortality | At day 90 after ICU admission
Time to S. aureus ICU pneumonia | day of ICU admission until ICU discharge (on average 7 days after ICU admission)
Time to P. aeruginosa ICU pneumonia | day of ICU admission until ICU discharge (on average 7 days after ICU admission)
Time to all cause ICU pneumonia | day of ICU admission until ICU discharge (on average 7 days after ICU admission)
Time to all cause ICU bacteremia | day of ICU admission until ICU discharge (on average 7 days after ICU admission)
Time to death of any cause | day of ICU admission until day 90 or ICU discharge, whichever comes first

OTHER OUTCOMES:
Magnitude of healthcare utilization as measured by: a. Duration of ICU stay including readmissions | day of ICU admission until day 30 after ICU discharge
Magnitude of healthcare utilization as measured by: b. Days on mechanical ventilation | day of ICU admission until ICU discharge (on average 9 days after ICU admission)
Magnitude of healthcare utilization as measured by: c. Days of antibiotic usage | day of ICU admission until ICU discharge (on average 9 days after ICU admission)
Magnitude of healthcare utilization as measured by: d. Duration of hospital stay, including readmissions | day of ICU admission until ICU discharge (on average 9 days after ICU admission)
Incidence of S. aureus colonization | from day of ICU admission until onset of ICU pneumonia (on average 7 days after ICU admission)
Incidence of P. aeruginosa colonization | from day of ICU admission until onset of ICU pneumonia (on average 7 days after ICU admission)

CONTACTS AND LOCATIONS:
Overall Officials: Jan A.J.W. Kluytmans, Prof., Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Engelen TSR, Reijnders TDY, Paling FP, Bonten MJM, Timbermont L, Malhotra-Kumar S, Kluytmans JAJW, Peters-Sengers H, van der Poll T; ASPIRE-I. C. U. Study Team. Plasma protein biomarkers reflective of the host response in patients developing Intensive Care Unit-acquired pneumonia. Crit Care. 2023 Jul 6;27(1):269. doi: 10.1186/s13054-023-04536-0. PMID 37415223
- [Derived] Paling FP, Troeman DPR, Wolkewitz M, Kalyani R, Prins DR, Weber S, Lammens C, Timbermont L, Goossens H, Malhotra-Kumar S, Sifakis F, Bonten MJM, Kluytmans JAJW. Rationale and design of ASPIRE-ICU: a prospective cohort study on the incidence and predictors of Staphylococcus aureus and Pseudomonas aeruginosa pneumonia in the ICU. BMC Infect Dis. 2017 Sep 25;17(1):643. doi: 10.1186/s12879-017-2739-4. PMID 28946849
- See also: Related Info — http://www.combacte.com